CLINICAL TRIAL: NCT06832332
Title: Midwifery Students' Experiences and Opinions on Alternative Birthing Positions in the Second Stage of Labor
Brief Title: Alternative Birth Positions During the Second Stage
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Mine Gokduman Keles, RESPONSIBLE RESEARCHER_ PhD midwife, Burdur Mehmet Akif Ersoy University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MAKÜ Unive
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Simulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- INTERVENTION 1 (Other)
  Interventions: Behavioral: alternative birthing positions
- Control Group (Active Comparator)
  Interventions: Behavioral: alternative birthing positions

INTERVENTIONS:
Behavioral: alternative birthing positions — In this stage, students will be given a simulated breech birth with alternative birth positions as opposed to the traditional position in the second stage of labor.

SUMMARY:
Simulation training provided before clinical practice at many universities helps students feel confident and well prepared for the clinical environment. Simulation-based learning not only improves professional competence in midwifery educators but also equips and empowers midwifery students in practice. In undergraduate midwifery education, students are provided obstetric skills training on electronic fetal monitoring (EFM), delivery management, shoulder dystocia, postpartum hemorrhage, breech delivery, umbilical cord prolapse and perineal repair (incision and episiotomy). It has been determined that simulation-based training positively affects the perceived readiness of the participants. It is emphasized that health personnel should be encouraged to freely choose birth positions and be informed about the risks and benefits of upright and supine positions. This study will be conducted to evaluate the effect of midwifery students' use of alternative birth positions in the second stage of labor on students' anxiety, self-efficacy, skill and knowledge levels.

ELIGIBILITY:
Inclusion Criteria:

* Continuing their third year in the 2024-2025 Spring semester,
* Students who have passed the normal birth management course

Exclusion Criteria:

* Students who fail the normal birth management course

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Childbirth Skills Self-Efficacy Scale | 1 HOUR